CLINICAL TRIAL: NCT01833962
Title: A Retrospective Study of Actifuse Synthetic Bone Graft Versus Other Bone Graft Substitutes in Patients Requiring Lumbar Fusion
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: OrthoGeorgia (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 001-3708
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Lumbar Fusion
Keywords: Lumbar fusion rates; Actifuse synthetic bone graft; Baxter Healthcare; Other synthetic bone graft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Actifuse: Patients who recieved Actifuse synthetic bone brafting material

SUMMARY:
The purpose of this study is to assess fusion status in patients who underwent spinal fusion with Actifuse synthetic bone graft versus other bone graft material (including autograft) in achieving lumbar spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* Any patient 18 years of age or older
* Patients with a minimum follow up of 1 year
* Patients who have previously undergone TLIF, PLIF,PLF, XLIF procedures

Exclusion Criteria:

* Patients under the age of 18
* Any patient with less than 1 year of follow up history at the time of first data analysis
* Any patient that the primary investigator deems as an unfit candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All study patients will be extracted from our current patient population. A total of 50 patients treated with Actifuse and 50 patients treated with other synthetic bone grafting substitutes
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Achievement of fusion prior to or at 12 months postoperatively | 6 - 12 months year

CONTACTS AND LOCATIONS:
Overall Officials: William B Dasher, MD, Principal Investigator — Physician
Locations (1):
- OrthoGeorgia, Macon, Georgia, United States

REFERENCES:
- See also: Related Info — http://www.orthoga.org